CLINICAL TRIAL: NCT02290145
Title: Cyclin D1 Based TPF(Docetaxel, Cisplatin and 5-fluorouracil) Induction Chemotherapy for OSCC(Oral Squamous Cell Carcinoma) Patients at cN2(Clinical Node 2) Stage: a Phase II Randomized Controlled Trial
Brief Title: Cyclin D1 Based TPF Induction Chemotherapy for Oral Squamous Cell Carcinoma Patients at Clinical N2 Stage
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Lai-ping Zhong, Professor,PHD,DDS,MD, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDSCAN
Record Dates: First submitted 2014-10-22; First posted 2014-11-13 (Estimated); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Mouth Neoplasms; Carcinoma, Squamous Cell
Keywords: docetaxel, cisplatin, 5-FU, cyclinD1
MeSH Terms: conditions — Mouth Neoplasms; Carcinoma, Squamous Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TPF group (Experimental): TPF induction chemotherapy followed with surgery and post-operative radiotherapy docetaxel 75mg/m2 cisplatin 75 mg/m2 5-Fu 750 mg/m2/day
  Interventions: Drug: TPF group; Procedure: surgery group; Radiation: Post-operative radiotherapy
- surgery group (Other): surgery with post-operative radiotherapy
  Interventions: Procedure: surgery group; Radiation: Post-operative radiotherapy

INTERVENTIONS:
Drug: TPF group — The patients in the experimental group received the TPF induction chemotherapy for 2 cycles followed by radical surgery and post-operative radiotherapy.
  docetaxel:75mg/m2 cisplatin：75 mg/m2 5-Fu：750 mg/m2/day
  Other Names: TPF protocol group
  Arms: TPF group
Procedure: surgery group — The patients in the control group received the radical surgery and post-operative radiotherapy.
Radiation: Post-operative radiotherapy — Radiotherapy was arranged 4 to 6 weeks after surgery. Routine external beam radiotherapy, such as conformal or intensity modulated radiotherapy was performed, and the dose was 1.8-2 Gy/day, 5 days/week for 6 weeks, and totally 54-60 Gy.

SUMMARY:
The purpose of this study is to To confirm the predictive value of CCND1 for TPF induction in cN2 patients with OSCC

DETAILED DESCRIPTION:
Induction chemotherapy is regarded as an effective way to reduce or downgrade the locally advanced or aggressive cancers, and to improve the chance of eradication of the locoregional lesions by radical surgery and/or radiotherapy. However, there are still debates on the clinical value of induction chemotherapy for patients with advanced and resectable oral squamous cell carcinoma. A prospective, open label, parallel, interventional, randomized control trial on TPF induction chemotherapy indicate there is no difference in overall survival, disease free survival, local regional recurrence free survival and metastasis free survival between experimental group and control group, however, the subgroup analysis proves that the induction chemotherapy of TPF protocol could benefit the patients with cyclinD1 high expression and cN2 locally advanced oral squamous cell carcinoma. （Zhong et al, Randomized Phase III Trial of Induction Chemotherapy With Docetaxel, Cisplatin, and Fluorouracil Followed by Surgery Versus Up-Front Surgery in Locally Advanced Resectable Oral Squamous Cell Carcinoma, J Clin Oncol 2013）The previous study was registered at ClinicalTrials.gov website with NCT01542931 identification number.This prospective, interventional, randomized control trial was to evaluate the TPF induction chemotherapy have a better effects in the cyclin D1 high expression and cN2 patients with locally advanced and resectable OSCC. The patients would receive TPF induction chemotherapy followed by radical surgery and post-operative radiotherapy (the experimental group) or radical surgery and post-operative radiotherapy (the control group). The primary endpoint is overall survival and the second endpoint is local control and distant control.The study had a power of 80% on the basis of an assumed 2-year survival rate of 67% in the experiment group and 25% in the control group, with use of a two-sided log-rank test at a level of significance of 0.05. The recruitment period would be 2 years, and the follow-up period would be 2 years, and 15% of patients would drop out early or be lost to follow-up. A maximum of 24 patients per group were to be recruited with stplan 4.5 software calculation. （Department of Biostatics, MD Anderson Cancer Center, University of Texas，USA）The patients in the experimental group received the TPF induction chemotherapy for 2 cycles followed by radical surgery and post-operative radiotherapy. The palpable edges of the primary lesion (both the longest and shortest axis) were marked before induction chemotherapy by at least four points, which were 0.5cm away. The patients in the control group received the radical surgery and post-operative radiotherapy.

Induction chemotherapy: For the patients who were randomly assigned to receive TPF induction chemotherapy, peripherally inserted central catheter was firstly inserted before intravenous infusion, docetaxel(at a dose of 75mg/m2 of body surface area) was administered as a 2-hour intravenous infusion, followed by intravenous cisplatin(75 mg/m2), administered during a period of 2 to 3 hours. Then, 5-Fu(5 - Fluorouracil) (750 mg/m2/day) was administered as a 120-hour continuous intravenous infusion for 5 days. Induction chemotherapy was given every 3 weeks for 2 cycles, unless there was disease progression, unacceptable toxic effects, or withdrawal of consent by the patients. Dexamethasone was given before docetaxel infusion to prevent docetaxel-related hypersensitivity reactions, skin toxic effects, and fluid retention; prophylactic antibiotics were also given starting on day 5 of each cycle for 3 days. Hydration with diuretic and antiemetic treatment was also performed. Primary prophylaxis with recombinant granulocyte colony-stimulating factor was not suggested. Chemotherapy dose reductions were allowed for grade 3/4 toxicities occurring after cycle 1: 25% and 50% dose reductions of the three chemotherapy agents were suggested for grade 3 and grade 4 hematologic toxicities or gastrointestinal toxicities, respectively; 25% and 50% cisplatin dose reductions were suggested for grade 3 and grade 4 renal toxicities, respectively. Surgery was performed at least 2 weeks after completion of induction chemotherapy.

Surgery: Radical resection of the primary lesion and full neck dissection(functional or radical) with proper reconstruction(pedicle or free flap) were performed. The safety margins of the primary lesion were 1.0-1.5cm far away from the palpable margins of the lesion; for patients who received induction chemotherapy, the safety margins were 1.0cm away from the marks that were placed before induction chemotherapy, to ensure the same extent surgery in both arms. Frozen sections during surgery were performed to confirm adequate margins.

Post-operative radiotherapy: Radiotherapy was arranged 4 to 6 weeks after surgery. Routine external beam radiotherapy, such as conformal or intensity modulated radiotherapy was performed, and the dose was 1.8-2 Gy/day, 5 days/week for 6 weeks, and totally 54-60 Gy, in the patient with high risk features, such as positive surgical margin, extra capsular nodal spread, vascular embolism, concurrent chemotherapy with cisplatin 80mg/m2 was suggested.

A complete medical history was obtained and tumor assessment was performed at baseline. Clinical tumor response was assessed by clinical evaluation and imaging study and was characterized according to the criteria of response evaluation criteria in solid tumors (version 1.1) before surgery. Post-operative pathologic response was assessed by post-operative pathologic examination as good and bad response. A good response was defined as absence of any tumor cells (pathologic complete response) or presence of scattered foci of a few tumor cells (minimal residual disease with <10% viable tumor cells); otherwise, a bad pathologic response was defined. Toxic effects were assessed weekly during and after completion of induction chemotherapy and radiotherapy according to the common terminology criteria for adverse events (version 3.0).

Overall survival was calculated from the date of randomization to the date of death; disease free survival was calculated from the date of randomization to tumor recurrence or distant metastasis or death from any cause; locoregional recurrence/distant metastasis free survival was calculated from the date of randomization to locoregional recurrence/distant metastasis of tumor or death from any cause. Time to locoregional recurrence/distant metastasis was calculated from the date of finishing treatment to tumor locoregional recurrence/distant metastasis. Patients were monitored by every three months in the first two years, every six months in the next 2 years, and once a year thereafter until death or data censoring.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 to 75 years old.
* Sex: both males and females.
* Karnofsky performance status (KPS) >60.
* Histological biopsy confirming squamous cell carcinoma of the oral cavity (tongue, gingiva, buccal mucosa, floor of mouth, palate, and retromolar region).
* Cyclin D1 high expression
* Clinical stage III/IVA (T1-2, N2, M0 or T3-4, N2, M0, UICC[International Union Against Cancer] 2002) with resectable lesions.
* Adequate hematologic function: white blood cell >3,000/mm3, hemoglobin>8g/L, platelet count>80,000/mm3.
* Hepatic function: ALAT(alanine aminotransferase)/ASAT(aspartate transaminase) <2.5 times the upper limit of normal (ULN), bilirubin <1.5 times ULN.
* Renal function: serum creatinine <1.5 times ULN.
* Written informed consent

Exclusion Criteria:

* Evidence of distant metastatic disease and other cancers.
* Surgical procedure of the primary tumors or lymph nodes (except diagnostic biopsy).
* Previous radiotherapy or chemotherapy.
* Other previous malignancies within 5 years.
* Can not tolerate the treatment protocol with systematic diseases such as history of severe pulmonary or cardiac diseases.
* Legal incapacity or limited legal capacity.
* Creatinine clearance <30ml/min.
* Pregnancy (confirmed by serum or urine β-HCG) or lactation period.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2016-12; Primary Completion 2024-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
overall survival rate as a measure by the numbers of living patients | 2 year

SECONDARY OUTCOMES:
disease free survival as a measure by the number of patients without recurrence or death | 2 year
local recurrence free survival as a measure by the number of patients without recurrence | 2 year
distant metastasis free survival as a measure by the number of patients without metastasis | 2 year

CONTACTS AND LOCATIONS:
Locations (1):
- Ninth People's Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China